CLINICAL TRIAL: NCT00325104
Title: Cinacalcet Actions in Familial Primary Hyperparathyroidism
Brief Title: Cinacalcet to Treat Familial Primary Hyperparathyroidism
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Purpose: Treatment
Other Study IDs: 060163; 06-DK-0163
Record Dates: First submitted 2006-05-11; First posted 2006-05-12 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2007-03-31

CONDITIONS: Hypercalcemia; Familial Primary Hyperparathyroidism
Keywords: Multiple Endocrine Neoplasia; Gastrinoma; Prolacinoma; Medullary Thyroid Cancer; Insulinoma; MEN1; MEN2A; Familial Primary Hyperparathytoidism
MeSH Terms: conditions — Hypercalcemia; Hyperparathyroidism 1; Multiple Endocrine Neoplasia; Gastrinoma; Carcinoma, Medullary; Insulinoma; Multiple Endocrine Neoplasia Type 2a

INTERVENTIONS:
Procedure: Parathyroid hormone testing
Procedure: Serum calcium testing

SUMMARY:
This study will evaluate the benefits and side effects of a new medication called Cinacalcet for treating patients with primary hyperparathyroidism associated with multiple endocrine neoplasia type 1 (MEN1) or type 2A (MEN2A). Patients with primary hyperparathyroidism have elevated levels of blood calcium caused by too much parathyroid hormone released by one or more parathyroid tumors. The parathyroids are small glands located in the neck. Most cases of primary hyperparathyroidism are due to a single overactive parathyroid gland, but in MEN1 and MEN2A, several glands are overgrown and overactive. Cinacalcet decreases the secretion of parathyroid hormone.

Patients 18 years of age and older with primary hyperparathyroidism and MEN1 or MEN2A and who are not candidates for parathyroid surgery may be eligible for this study.

Participants are admitted to the Clinical Center for 1 week blood and urine tests and imaging studies, and initiation of Cinacalcet treatment. They take the drug by mouth and have daily blood tests until the dosage required to achieve normal blood calcium levels is determined. Patients return to the hospital 2 weeks later for 1 week to evaluate the response to the drug and make any necessary adjustments. Treatment may continue for as long as 1 year with 1-week admissions every 3 months to monitor the benefits and side effects of Cinacalcet. Evaluations may include the following:

* Blood and urine analyses.
* Measurement of gastric acid secretion. For this test, a soft plastic tube is inserted into the nose or mouth and then swallowed and then gently removed about an hour later.
* Injections of secretin, calcium and arginine into a vein and collection of blood samples to measure the responding increase in levels of gastrin, calcitonin and insulin, respectively. These tests are used to diagnose and monitor hormone secretion from endocrine tumors and are used in this study to assess the response to Cinacalcet treatment.
* Radioisotope test to evaluate tumors of the endocrine organs. A radioactive substance injected into a vein is taken up by the endocrine tissue and the concentrated radioactivity is measured.
* Imaging tests, such as MRI and CT, to detect or follow growing tumors in the pituitary, neck, and abdomen. CT is a special type of x-ray machine that visualizes tissues, such as thyroid or parathyroid tumors. MRI uses a magnetic field and radio waves to obtain pictures of different tissues in the head, neck and abdomen.
* DEXA scan to assess bone density. This test uses standard low-intensity x-rays.

DETAILED DESCRIPTION:
This study will evaluate safety and efficacy of short- and long-term Cinacalcet in treatment of hypercalcemia of familial primary hyperparathyroidism. The study population will include patients with primary hyperparathyroidism caused by multiple endocrine neoplasia type 1 or type 2A. This is a prospective unblinded pilot study, where each patient will serve as his/her own control. It will include 6 one-week-long admissions, over a 1 year period. Main measurements will be tests of hyperparathyroidism such as parathyroid hormone and serum calcium as well as tests of nonparathyroid tumors. The latter tests may include hormones released by the tumors and images of the tumors.

ELIGIBILITY:
* INCLUSION CRITERIA:

Criteria for inclusion

1. Patients with primary hyperparathyroidism associated with MEN1 or 2A syndrome and no indications for current surgical interventions.
2. For initial pilot study, 15-20 patients with MEN1 syndrome and biochemical evidence of hyperparathyroidism will be included.
3. For initial pilot study, 5-10 patients with MEN2A syndrome and biochemical evidence of hyperparathyroidism will be included. Each MEN2A case must have residual MTC tumor.
4. In case of ZES, good acidity control with proton pump inhibitors (PPI), documented by basal acid output (BAO) of less than 10 mEq/h.
5. Willingness and legal ability to give informed consent.
6. MEN1, like MEN2A has a normal gender and ethnic distribution. These will be maintained, within the limits of a small number of subjects studied.

EXCLUSION CRITERIA:

Criteria for exclusion or removal

1. Age less than 18 years
2. Pregnancy
3. Creatinine greater than 1.4
4. SGOT or SGPT greater than twice normal
5. Indications for current surgery:

   1. Hyperparathyroidism

      * Albumin-adjusted serum calcium level higher than 3.0 mmol/L (12.0 mg/dL)
      * Kidney stones
      * Significant PTH-induced bone disease
      * Age below 50 is not considered as absolute indication for parathyroid surgery herein
   2. Enteropancreatic neuroendocrine neoplasia

      * Single lesion meeting criteria for surgery
      * Need for debulking surgery for obstructive or other complications
      * Acute abdominal complications of any kind
      * Inability of control on PPI in case of ZES
6. Chemotherapy within last 6 months
7. Lactating females
8. Patients with contraindications for MRI study, including pacemakers, vascular clips, implants, foreign bodies etc., as per NIH-MRI Safety Guideline.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25
Dates: Start 2006-05-09; Study Completion 2007-03-31

CONTACTS AND LOCATIONS:
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Rizzoli R, Green J 3rd, Marx SJ. Primary hyperparathyroidism in familial multiple endocrine neoplasia type I. Long-term follow-up of serum calcium levels after parathyroidectomy. Am J Med. 1985 Mar;78(3):467-74. doi: 10.1016/0002-9343(85)90340-7. PMID 2858157